CLINICAL TRIAL: NCT03613857
Title: Combined Effect of Diabetes and cyp2c19 Polymorphism on Clopidogrel VS Ticagrelor Antiplatelet Activity in Patients of Anterior ST Elevation Myocardial Infarction Undergoing Primary PCI
Brief Title: Effect of Diabetes and Hepatic Enzymes Mutation on Clopidogrel VS Ticagrelor Activity in Myocardial Infarction (MI) Patients Undergoing Primary Percutaneous Coronary Intervention (PCI)
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mina Wageh Mohareb, researcher at clinical pharmacology department cairo university, principal investigator, Cairo University
Other Study IDs: pharmacology department CU
Record Dates: First submitted 2018-07-29; First posted 2018-08-03 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — Clopidogrel; Ticagrelor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Blood samples.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Clopidogrel group: Anterior myocardial infarction patients undergoing percutaneous coronary intervention take loading dose 600 mg oral clopidogrel (plavix) tablets before the procedure.
  Interventions: Drug: Clopidogrel
- Ticagrelor group: Anterior myocardial infarction patients undergoing percutaneous coronary intervention take loading dose180 mg oral ticagrelor (brilique) tablets before the procedure.
  Interventions: Drug: Ticagrelor 90mg

INTERVENTIONS:
Drug: Clopidogrel — 8 tablets 75 mg clopidogrel loading dose before PCI
  Other Names: plavix
  Groups: Clopidogrel group
Drug: Ticagrelor 90mg — 2 tablets 90 mg brilique before PCI
  Other Names: brilique
  Groups: Ticagrelor group

SUMMARY:
In this study the combined effect of diabetes mellitus and cyp2c19 polymorphism on platelet aggregation inhibitory activity of the highest traditionally used loading dose 600 mg clopidogrel and ticagrelor 180 mg loading dose will be compared in acute coronary syndrome (ACS) patients undergoing PCI.

DETAILED DESCRIPTION:
Study subjects Inclusion criteria Diabetic patients (well-controlled type 2 diabetes mellitus) and non-diabetic patients with anterior ST-elevation and non-st elevation myocardial infarction undergoing PCI.

Exclusion criteria Patients who are with a family or personal history of bleeding. Patients with platelet count less than 100 x 103/ul. Patients with known hypersensitivity to clopidogrel or ticagrelor. Patients with serious bleeding tendency, history of intracranial hemorrhage, a sign of active bleeding, uncontrolled hypertension.

Patients with severe liver disorders

Methods The study will be conducted in the cardiac intensive care unit at Assiut educational hospital of cardiovascular diseases.

* diabetic and non-diabetic patients with ST-elevation and non-ST elevation myocardial infarction undergoing PCI will be enrolled in this study.
* At baseline, all patients will undergo full clinical examination and laboratory diagnostic tests. Current and previous medical history and medication history will be thoroughly investigated.

Recruited patients will be classified into two groups. One group will receive 600 mg loading dose clopidogrel before PCI and 75 mg daily maintenance dose. The other group of patients will receive 180 mg loading dose ticagrelor before PCI and 90 mg twice daily maintenance dose.

A blood sample of will be withdrawn from each patient to undergo genotypic testing using Real Time polymerase chain reaction (PCR) to detect polymorphism in the cyp2c19 enzyme.

* Clopidogrel and ticagrelor antiplatelet activity will be assessed by estimating the maximum platelet aggregation (MPA) using light transmittance platelet aggregometry and platelet reactivity index (PRI) using whole-blood vasodilator-stimulated phosphoprotein (VASP) measured by quantitative flow cytometry.
* All patients will be followed-up for at least three to six months month by clinic visits and phone calls to detect acute and subacute stent thrombosis, acute cardiac events, revascularization and cardiovascular death after PCI.

Study endpoints Acute stent thrombosis 24 hours after PCI and sub-acute stent thrombosis within 30 days after PCI, cardiovascular death, recurrent acute cardiac events, recurrent unstable anginal pain and hospitalization for cardiovascular diseases.

ELIGIBILITY:
Inclusion Criteria:

-Diabetic and non-diabetic patients with anterior ST-elevation and non-ST elevation myocardial infarction undergoing PCI.

Exclusion Criteria:

* Patients who are with a family or personal history of bleeding.
* Patients with platelet count less than 100 x 103/ul.
* Patients with known hypersensitivity to clopidogrel.
* Patients with serious bleeding tendency, history of intracranial hemorrhage, signs of active bleeding, uncontrolled hypertension.
* Patients with severe liver disorders

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic and non-diabetic patients with ST-elevation elevation and non-ST elevation myocardial infarction undergoing PCI.
Sampling Method: Non-Probability Sample
Enrollment: 1022 (Actual)
Dates: Start 2017-04-15 (Actual); Primary Completion 2018-07-28 (Actual); Study Completion 2018-07-28 (Actual)

PRIMARY OUTCOMES:
Acute and sub-acute stent thrombosis | up to one month after stent implantation
  stent thrombosis 24 hr to one month after stent implantation
Cardiovascular death | three to six months after PCI
  Death with cardiovascular etiology
Non-fatal myocardial infarction | three to six months after PCI
  Survival after hospital admission due to ST elevation or non-ST elevation myocardial infarction
Ischemic or hemorrhagic stroke | three to six monthes after PCI

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of pharmacy Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mohareb MW, AbdElghany M, Zaki HF, El-Abhar HS. Diabetes and CYP2C19 Polymorphism Synergistically Impair the Antiplatelet Activity of Clopidogrel Compared With Ticagrelor in Percutaneous Coronary Intervention-treated Acute Coronary Syndrome Patients. J Cardiovasc Pharmacol. 2020 Oct;76(4):478-488. doi: 10.1097/FJC.0000000000000881. PMID 32675750